CLINICAL TRIAL: NCT06957899
Title: Impact of Spinal Needle Gauge on Optic Nerve Sheath Diameter in Patients With Post-Dural Puncture Headache
Brief Title: Optic Nerve Sheath Diameter in Postspinal Headache
Acronym: PDPHPatients
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Nuran Akıncı Ekinci, MD, Specialist in Anesthesiology, Konya City Hospital
Other Study IDs: 2025/38
Record Dates: First submitted 2025-04-12; First posted 2025-05-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Post-Dural Puncture Headache
Keywords: Post-Dural Puncture Headache (PDPH); Intracranial Hypotension; Spinal Anesthesia Complication; Optic Nerve Sheath Diameter; Spinal Needle Gauge
MeSH Terms: conditions — Post-Dural Puncture Headache; Intracranial Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 25: Group 25G: Patients who underwent spinal anesthesia with a 25-gauge needle
- Group 27: Group 27G: Patients who underwent spinal anesthesia with a 27-gauge needle

SUMMARY:
This study aims to investigate the relationship between spinal needle size and optic nerve sheath diameter (ONSD) in patients who develop post-dural puncture headache (PDPH) after spinal anesthesia. ONSD is measured using ultrasound, which helps estimate changes in brain pressure. The study also examines whether the severity of headache is related to ONSD. Adult patients aged 18 to 75 years who develop PDPH will be included. This research will be conducted at Konya City Hospital and is expected to last for approximately six months.

DETAILED DESCRIPTION:
This prospective observational study investigates the relationship between spinal needle gauge and optic nerve sheath diameter (ONSD) in patients who develop post-dural puncture headache (PDPH) following spinal anesthesia. ONSD is measured using ultrasound as a non-invasive marker of intracranial pressure. The study also aims to evaluate the association between headache severity, assessed by the Visual Analog Scale (VAS), and ONSD values. Patients aged 18-75 years with PDPH will be included, and data on spinal needle gauge, ONSD, and VAS scores will be analyzed. The study is being conducted at a single tertiary care center and aims to contribute to understanding the physiopathology of PDPH and its relation to procedural factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with postdural puncture headache (PDPH)
* Male and female patients aged 18-75 years
* Patients classified as American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Presence of neurological or ophthalmological disorders
* History of head trauma within the past 6 months
* Hypertension
* Hepatic encephalopathy
* Renal failure
* Pregnancy
* History of chronic headache or migraine
* Refusal to participate
* Inability to obtain reliable optic nerve sheath diameter (ONSD) measurements
* Communication difficulties preventing assessment
* Incomplete or inaccessible medical records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 75 years who develop post-dural puncture headache (PDPH) following spinal anesthesia. All participants are evaluated and monitored at a tertiary care center and are classified as ASA physical status I to III.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) | Within 4 hours of anesthesia consultation for postoperative headache
  The primary outcome is the measurement of optic nerve sheath diameter (ONSD) via ocular ultrasound in patients who develop postoperative headache attributed to dural puncture. This non-invasive assessment is used to estimate intracranial pressure. The aim is to evaluate whether different spinal needle gauges affect ONSD measurements.

SECONDARY OUTCOMES:
Pain severity assessed by Visual Analog Scale (VAS) | Within 4 hours of anesthesia consultation for postoperative headache
  Pain severity will be scored using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain), during the anesthesia consultation conducted for postoperative headache. This measure will be compared with ONSD values.

OTHER OUTCOMES:
Spinal Needle Gauge | Retrieved from procedure documentation at the time of spinal anesthesia
  The gauge (diameter in G) of the spinal needle used for the neuraxial procedure will be extracted from anesthesia records. The goal is to assess whether the spinal needle size is associated with ONSD measurements in patients with postoperative headache.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran AKINCI EKİNCİ, Study Chair — Konya City Hospiital
Locations (1):
- Konya City Hospital, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang P, Zhou X, Sheng F, Wang X, Shi C, Feng W. Ultrasonic optic nerve sheath diameter can be used as a diagnostic measure after accidental dural puncture during cesarean section: a case report. BMC Anesthesiol. 2024 Jan 22;24(1):35. doi: 10.1186/s12871-024-02418-8. PMID 38254029
- [Background] Dubost C, Le Gouez A, Zetlaoui PJ, Benhamou D, Mercier FJ, Geeraerts T. Increase in optic nerve sheath diameter induced by epidural blood patch: a preliminary report. Br J Anaesth. 2011 Oct;107(4):627-30. doi: 10.1093/bja/aer186. Epub 2011 Jun 21. PMID 21693468